CLINICAL TRIAL: NCT03928379
Title: A Multiple-Ascending Dose Study in Patients With Type 2 Diabetes Mellitus to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3305677
Brief Title: A Study of LY3305677 in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17011; I8P-MC-OXAD (Other: Eli Lilly and Company); 2018-004779-11 (EudraCT Number)
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3305677 (Experimental): LY3305677 administered SC
  Interventions: Drug: LY3305677
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3305677 — Administered SC
  Arms: LY3305677
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about the safety and side effects of LY3305677 when it is given as an injection just under the skin to participants with type 2 diabetes. The study will last about 20 weeks for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Have Type II diabetes
* Body mass index (BMI) of 25-40 kilograms per square meter (kg/m²), inclusive
* Have a body weight of <150 kilograms (kg)
* Have clinical lab test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator; however, should have serum magnesium and potassium levels, along with lactate dehydrogenase, CK values within the normal range at screening and Day -2.

Exclusion Criteria:

* Have Type 1 diabetes or latent autoimmune diabetes in adults
* Have uncontrolled diabetes defined as an episode of ketoacidosis or hyperosmolar state requiring hospitalization for 6 months prior to screening
* Have had an episode of severe hypoglycemia, defined by the occurrence of neuroglycopenic symptoms requiring the assistance of another person for recovery, within 6 months prior to Visit 1
* Have an abnormal 12-lead electrocardiogram (ECG) at screening and/or Day -2 that, in the opinion of the investigator, increases the risks associated with participating in the study or may confound ECG data analysis
* Have poorly controlled hypertension at screening; or a change in antihypertensive medication within 30 days of screening
* Have an estimated glomerular filtration rate <45 milliliters per minute per 1.73 meters squared of body surface area (mL/min/1.73 m²)

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug | Baseline through 24 weeks
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3305677 | Baseline through 48 hours postdose
  PK: Cmax of LY3305677
PK: Area Under the Concentration-Time Curve (AUC) of LY3305677 | Baseline through 48 hours postdose
  PK: AUC of LY3305677
Pharmacodynamics (PD): Change from Baseline in Fasting Plasma Glucose | Baseline, through Week 16
  PD: Change from Baseline in Fasting Plasma Glucose
PD: Change from Baseline in Fasting Plasma Insulin | Baseline, through Week 16
  PD: Change from Baseline in Fasting Plasma Insulin

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No